CLINICAL TRIAL: NCT05316740
Title: Vaginal Microbiome and the Risk of Vulvovaginal Graft Versus Host Disease Following Hematopoietic Stem Cell Transplantation
Brief Title: Vaginal Microbiome and the Development of Vulvovaginal Graft Versus Host Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Rambam Health Care Campus (Other); Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0512-21-HMO
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Bone Marrow Transplant Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal samples will be collected for:
  1. Microbiome molecular analysis: aimed to determine whether changes in the vaginal bacterial microbiome precede or follow VV-GVHD.
  2. HPV presence.
  3. CMV presence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — Repeated clinical evaluation and sample collection

SUMMARY:
Allogeneic stem cell transplantation (also termed "bone marrow transplantation") involves transferring stem cells from a healthy person (the donor) to the patient, after high-intensity chemotherapy or radiation, given to destroy any remaining cancer cells in the body. When a transplant is successful, the donor stem cells replace the original cells in the bone marrow. It may provide the only long-term cure of the patient's disease. Of transplant-related complications, graft-versus-host disease (GVHD) is one of the most important complications. GVHD arises from donor immune cells, that identify the recipient's (the patien's) cells as foreign and attack them. Approximately half of women undergoing transplantation will experience GVHD involving the genitalia (i.e., the vulva and vagina), termed vulvovaginal GVHD (VV-GVHD). VV-GVHD may cause irreversible anatomical changes, including complete vaginal obliteration, and not surprisingly, it has a severe impact on patients' quality of life and sexual function. This complication is unpredictable and non-preventable by the usual immunosuppressive treatment given to patients. Frequent gynecological examinations and prolonged follow-up of transplanted women are needed, to allow early diagnosis and prevention of harmful results of VV-GVHD. This follow-up adds inconvenience and anxiety to the patients.

The suggested study aims to evaluate a possible association between vaginal microorganisms (the "microbiome") to the progress of VV-GVHD. Finding such association may allow prediction of VV-GVHD progress, a better understanding of the development of VV-GVHD and a potential to develop interventions for the treatment and prevention of VV-GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* Candidate for allogeneic stem cell transplantation
* Ability to sign an informed consent

Exclusion Criteria:

- Patient does not approve sample collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients planned for HSCT
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition | 2 years
  Characterization of the vaginal microbial community using shotgun analysis and16S rRNA sequencing
CMV presence | 2 years
  Evaluation of CMV in vaginal samples using PCR assay
Vulvovaginal graft vs host disease presence | 2 years
  Evaluation of presence of vulvovaginal GVHD by gynecologic examination, using the NIH classification system for chronic graft-versus-host disease

SECONDARY OUTCOMES:
HPV presence | 2 years
  Evaluation of HPV in vaginal samples

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev Sagie, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Jerusalem, Israel